CLINICAL TRIAL: NCT00080054
Title: Phase I Trial of Motexafin Gadolinium (MGd) in Combination With Temozolomide for Treatment of Malignant Gliomas
Brief Title: A Study of Motexafin Gadolinium and Temozolomide for the Treatment of Malignant Gliomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pharmacyclics LLC. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PCYC-0218
Record Dates: First submitted 2004-03-22; First posted 2004-03-23 (Estimated); Last update posted 2009-04-03 (Estimated); Status verified 2007-01

CONDITIONS: Glioma; Glioblastoma; Astrocytoma; Oligodendroglioma; Brain Neoplasm
Keywords: Malignant Glioma; Glioblastoma multiforme; GBM; Anaplastic astrocytoma; AA; Anaplastic oligodendroglioma; Anaplastic mixed glioma; Brain tumor; Brain neoplasm; Glioma
MeSH Terms: conditions — Glioma; Glioblastoma; Astrocytoma; Oligodendroglioma; Brain Neoplasms | interventions — motexafin gadolinium

INTERVENTIONS:
Drug: Motexafin Gadolinium Injection

SUMMARY:
The purpose of this study is to find out about the safety of adding the investigational drug motexafin gadolinium to a standard course of chemotherapy with temozolomide for patients with malignant glioma. Secondly, the study will determine how many patients will respond to this treatment.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Histologically confirmed diagnosis of malignant gliomas that requires systemic antineoplastic treatment. Malignant glioma is defined as any of the following: Glioblastoma multiforme (GBM); Anaplastic astrocytoma (AA); Anaplastic oligodendroglioma; Anaplastic mixed glioma; Glioma not otherwise specified (except low-grade glioma)
* ECOG performance status score of 0, 1, or 2
* Each patient must sign a study-specific informed consent form

Exclusion Criteria:

Laboratory values of:

* Absolute neutrophil count < 2000/µL
* Platelet count < 100,000/µL
* AST or ALT > 2 x the upper limit of normal (ULN)
* Alkaline phosphatase > 5 x ULN
* Bilirubin > 2 x ULN
* Creatinine > 2.0 mg/µL

and

* Plan to use any additional cancer therapy (e.g., systemic, radiation, surgery) during the study period
* Women who are pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24

CONTACTS AND LOCATIONS:
Locations (1):
- Barrow Neurological Institute, Phoenix, Arizona, United States

REFERENCES:
- See also: Related Info — http://www.braintumor.org
- See also: Related Info — http://www.pcyc.com